CLINICAL TRIAL: NCT03569085
Title: Effect of Inhalational Anesthetics on Myocardial Deformation Indices - A Dose-Response Cross-over Study
Brief Title: Inhaled Anesthetics and Myocardial Strain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kathirvel Subramaniam (Other)
Responsible Party: Sponsor-Investigator, Kathirvel Subramaniam, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PRO17080624
Record Dates: First submitted 2018-06-01; First posted 2018-06-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Intervention Model Description: Same patients will receive two different arms/interventions and compared
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sevoflurane then isoflurane (Experimental)
  Interventions: Drug: Sevoflurane; Drug: Isoflurane

INTERVENTIONS:
Drug: Sevoflurane — The patient will receive Sevoflurane in incremental doses titrated to obtain end-tidal minimum alveolar concentration (MAC) of 0.5, 1.0, and 1.5.
Drug: Isoflurane — The patient will receive isoflurane in incremental doses titrated to obtain end-tidal minimum alveolar concentration (MAC) of 0.5, 1.0, and 1.5.

SUMMARY:
Speckle tracking imaging measuring software will be used for offline analysis of transesophageal echocardiogram (TEE) -acquired images of the left ventricle(LV) in four chambers(4C), two chambers (2C) and long axis (LAX) views to calculate global longitudinal strain (GLS) of LV for comparisons between sevoflurane and isoflurane at the same minimum alveolar concentration ( MAC) levels.

DETAILED DESCRIPTION:
The primary research activity will be: baseline transthoracic echocardiogram (TTE) views taken upon the patient entering the operating room by one of the cardiothoracic anesthesiology fellows or attendings, TEE views taken by the echocardiography fellow or attending in the mid-esophageal 4C, 2C and LAX views once the patient has reached sevoflurane end-tidal minimum alveolar concentration (MAC) of 0.5, 1.0, and 1.5. Following this, sevoflurane will be changed to isoflurane and wait till complete washout of sevoflurane (i.e. end-tidal sevoflurane concentration reaches zero). Isoflurane concentration will be adjusted according to bispectral index and hemodynamics to maintain anesthesia during this period. Once complete sevoflurane wash-out has been achieved, isoflurane concentration will be adjusted and repeat images taken at the 0.5, 1.0, and 1.5 MAC values.

Investigators will establish stability at each MAC level (0.5, 1.0 and 1.5) for 5 minutes before obtaining TEE images. The whole study is done during pre- cardiopulmonary bypass(CPB) period while surgeon spending time dissecting internal mammary artery or other parts of surgical dissection before heparinization. The entire study duration will be a maximum of 35-40 minutes and this will not prolong the operating time. The adjustment of the anesthetic will be performed by the cardiac anesthesiology fellow or senior resident involved in this research along with the faculty officially performing the case. All images will be acquired prior to the initiation of cardiopulmonary bypass by the echocardiography rotating resident or research resident, cardiac anesthesiology fellow or cardiac anesthesiology attending anesthesiologist (all received extensive training in TEE to obtain those required images). Following the completion of the case and the uploading of images to a central echocardiography server, one of the study personnel will perform analysis of the images in the anesthesiology offices on a computer with post-processing software to determine strain.

MAC up to 1.5 is very well tolerated in cardiac surgical patients and is routinely used to achieve hemodynamic conditions during surgery. Use of vasopressor and inotrope to allow maintain depth of anesthesia with inhalation anesthesia agents is also routine in cardiac surgical patients and not in any way different from routine clinical care.

Hemodynamic information (heart rate, blood pressure, central venous pressure, cardiac index or pulmonary artery pressure) will be obtained after stabilization with each MAC and will be recorded immediately or extracted from the electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

Adult Patients (> 18 years of age) undergoing cardiovascular surgery at University of Pittsburgh Medical Center (UPMC) Presbyterian hospital.

Exclusion Criteria:

Inability to comprehend and understand the study, Pregnancy Malignant hyperthermia Acute cardiogenic shock and ongoing chest pain Permanent pacemaker with pacemaker dependency Abnormal cardiac rhythms ( e.g. atrial fibrillation) Contraindications to TEE examination such as recent esophageal surgery, esophageal cancer/stricture The use of anesthesia maintenance with intravenous anesthesia drugs such as propofol infusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Global longitudinal strain of myocardium, unitless (Comparison between two inhalational anesthetics, isoflurane and sevoflurane) | Intraoperative period during cardiac surgery before initiation of cardiopulmonary bypass
  Global longitudinal Strain measures changes in longitudinal length of myocardium and is a unitless measure. TEE images will be taken during surgery, stored on central echocardiography server, then analyzed offline using a special software to calculate global longitudinal strain (GLS). GLS of LV will then be compared between isoflurane and sevoflurane at the same MAC concentrations.

SECONDARY OUTCOMES:
Global longitudinal strain of myocardium, unitless (Dose dependent effect of sevoflurane) | Intraoperative period during cardiac surgery before initiation of cardiopulmonary bypass
  Global longitudinal Strain measures changes in longitudinal length of myocardium and is a unitless measure. TEE images will be taken during surgery, stored on central echocardiography server, then analyzed offline using a special software to calculate global longitudinal strain (GLS). GLS of LV will then be compared at increasing MAC of sevoflurane.
Global longitudinal strain of myocardium, unitless (Dose dependent effect of isoflurane) | Intraoperative period during cardiac surgery before initiation of cardiopulmonary bypass
  Global longitudinal Strain measures changes in longitudinal length of myocardium and is a unitless measure. TEE images will be taken during surgery, stored on central echocardiography server, then analyzed offline using a special software to calculate global longitudinal strain (GLS). GLS of LV will then be compared at increasing MAC of isoflurane.

CONTACTS AND LOCATIONS:
Overall Officials: Kathirvel Subramaniam, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States